CLINICAL TRIAL: NCT04842162
Title: Study Evaluating Near-infrared Imaging Coupled With Indocyanine Green for Intraoperative Control of Resection Margins in ENT Surgery
Acronym: MAGNOLIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-002442-20; 2019/2886 (Other: CSET number)
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized bicentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with head and neck cancer (Experimental)
  Interventions: Drug: indocyanine green

INTERVENTIONS:
Drug: indocyanine green — indocyanine green (INFRACYANINE© 25mg/10mL).

SUMMARY:
Assess the sensitivity of real-time near-infrared fluorescence imaging to detect microscopic residual disease in the operating room after a complete macroscopic surgical resection of head and neck cancers

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* ECOG performance status 0-2
* Histological confirmation of squamous cell carcinoma
* Locating the primary tumour in the oral cavity or oropharynx
* Disease operable for complete resection
* Serum or urinary pregnancy test (as per centre practices) negative within 14 days prior to systemic indocyanin green injection (pre-operative visit), for women of childbearing age
* Patient information and signed free and informed consent
* Patient affiliated with a social security scheme or beneficiary of a similar scheme.
* The patient must understand, sign and date the consent form prior to any protocol-specific procedures. The patient must be able and willing to comply with the study visits and procedures described in the protocol

Exclusion Criteria:

* Severe medical co-morbidities or contraindications to surgery
* Primary tumour not operable
* History of head and neck cancer in the past 5 years
* History of radiation for head and neck cancer
* Metastatic cancer
* Tumours with necrosis ranges in pre-operative imaging
* History of invasive cancer unless there has been no recurrence for more than 5 years with an exception for non-melanoma skin cancers.
* Pregnant or nursing woman
* Allergy or hypersensitivity to the product being administered (its active substance or other ingredients), iodized products or crustaceans.
* Hyperthyroidism, thyroid adenoma, unifocal, multifocal or multinodular goiter of autoimmune origin.
* Documented coronary artery disease
* Advanced renal failure (creatinine > 1.5mg/dL).
* Within 2 weeks prior to inclusion, concomitant medication that reduces or increases extinction of GI (i.e. anticonvulsants, haloperidol and Heparin).
* Patient under guardianship or curatorship or deprived of liberty by judicial or administrative decision or patient unable to give consent.
* Patients unable to undergo medical follow-up of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Near Infrared Fluorescence Imaging | at surgery
  Sensitivity of real-time near-infrared fluorescence imaging to detect microscopic residual disease in the operating room after complete macroscopic surgical resection.
  For the calculation of the sensitivity, for each operating room we consider the first section and the last section in which the pathological analysis confirms the presence of microscopic residual disease. Patients for whom near-infrared fluorescence imaging detects disease are classified as true positives (TP). Sensitivity is defined as the number of TP divided by the total number of patients N.

CONTACTS AND LOCATIONS:
Locations (2):
- Institut Jules Bordet, Anderlecht, Belgium
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided